CLINICAL TRIAL: NCT01825772
Title: Clinical and Radiographic Outcomes of Dental Implant Therapy
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Social Insurance Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: Jan1
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Peri-Implantitis
Keywords: Cross-Sectional Studies; Prevalence; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
900 subjects having received dental implants 9-10 years ago are invited for a clinical and radiographic examination. The individuals were randomly selected from the National Health Insurance data register in Sweden.

The clinical and radiographic examination of the 900 selected subjects will include assessments of implant loss, loss of prosthesis and technical / biological complications.

Biological complications will be assessed from the findings in the clinical and radiographic examinations. Thus, signs of pathology in peri-implant tissues, probing pocket depth (PPD) and bleeding/pus on probing (BoP) will be recorded. Marginal bone loss and other findings in radiographs will also be evaluated.

The prevalence, extent and severity of peri-implantitis will hereby be determined. Patient-centered outcomes will also be obtained.

ELIGIBILITY:
A questionnaire was distributed to the 4716 identified subjects. 3827 questionnaires (81.15%) were returned and, hence, included in the analysis.

From the sample of 3827 patients who responded to the questionnaire, 3107 (81.19%) gave their consent for access of patient files/records.

Patient files/records of 2780 individuals could be collected from the treating dentists (89.48%). Out of the 2780, 900 individuals were selected by random sampling, stratifying only for the two age groups.

Inclusion Criteria:

* Having received implants within the Swedish insurance system in 2003/2004.
* Being in one of the two age groups in 2003: 65-75 years and 45 - 55 years.
* Having answered the initial questionnaire
* Treating dentist provided patient files/records

Exclusion Criteria:

- Having died during the study period (collection of questionnaire and patient files/records)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The register of the Swedish Social Insurance Agency was searched for subjects scheduled for treatment with dental implants in 2003/2004. In a first group, subjects between 65 and 75 years old in 2003 were identified and from this pool of about 23.000 individuals, 3.000 subjects were randomly selected. In a second group, all subjects in the age of 45-60 years were identified (n=1716)from the same register. Thus, the total study population in the present project included 4716 subjects.
Sampling Method: Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Peri-implantitis | 9-10 years following implant installation
  All subjects were provided with dental implants in 2003/2004. The clinical and radiographic examinations will be carried out in 2013.

SECONDARY OUTCOMES:
Implant loss | 9-10 years after having received dental implants

OTHER OUTCOMES:
Technical complications | 9-10 years after receiving dental implants
  Technical complications relating to implant components or the prosthetic reconstruction are recorded. Recorded complications are (i) acrylic/porcelain fractures, (ii) screw-loosening and decementation, (iii) abutment screw loosening or fractures and (i) implant fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Tord Berglundh, Professor, Study Director — Göteborg University; Jan Derks, PhD Student, Principal Investigator — Göteborg University
Locations (1):
- Department of Periodontology, Institute of Odontology, Gothenburg, Sweden

REFERENCES:
- [Background] Fransson C, Lekholm U, Jemt T, Berglundh T. Prevalence of subjects with progressive bone loss at implants. Clin Oral Implants Res. 2005 Aug;16(4):440-6. doi: 10.1111/j.1600-0501.2005.01137.x. PMID 16117768
- [Background] Tomasi C, Derks J. Clinical research of peri-implant diseases--quality of reporting, case definitions and methods to study incidence, prevalence and risk factors of peri-implant diseases. J Clin Periodontol. 2012 Feb;39 Suppl 12:207-23. doi: 10.1111/j.1600-051X.2011.01831.x. PMID 22533958
- [Background] Berglundh T, Persson L, Klinge B. A systematic review of the incidence of biological and technical complications in implant dentistry reported in prospective longitudinal studies of at least 5 years. J Clin Periodontol. 2002;29 Suppl 3:197-212; discussion 232-3. doi: 10.1034/j.1600-051x.29.s3.12.x. PMID 12787220
- [Derived] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Peri-implantitis - onset and pattern of progression. J Clin Periodontol. 2016 Apr;43(4):383-8. doi: 10.1111/jcpe.12535. Epub 2016 Mar 29. PMID 26900869
- [Derived] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Derived] Derks J, Hakansson J, Wennstrom JL, Tomasi C, Larsson M, Berglundh T. Effectiveness of implant therapy analyzed in a Swedish population: early and late implant loss. J Dent Res. 2015 Mar;94(3 Suppl):44S-51S. doi: 10.1177/0022034514563077. Epub 2014 Dec 11. PMID 25503901